CLINICAL TRIAL: NCT02520362
Title: Denosumab Global Safety Assessment Among Women With Postmenopausal Osteoporosis (PMO), Men With Osteoporosis, and Men and Women Who Receive Prolia With Glucocorticoid Exposure in Multiple Observational Databases
Brief Title: Denosumab Safety Assessment in Multiple Observational Databases
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Collaborators: Aarhus University Hospital (Other); Optum, Inc. (Industry); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: 20090522
Record Dates: First submitted 2015-05-07; First posted 2015-08-11 (Estimated); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Denosumab; Diphosphonates

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Postmenopausal Women: Postmenopausal Women
- Women with post menopausal osteoporosis: Women with post menopausal osteoporosis
  Interventions: Drug: denosumab; Drug: bisphosphonate
- Prolia for unapproved indications: Patients who receive Prolia for unapproved indications
  Interventions: Drug: denosumab
- Men with osteoporosis: Men with osteoporosis treated with denosumab
  Interventions: Drug: denosumab
- Men and women who receive Prolia with Glucocorticoid exposure: Drug: denosumab subcutaneous injection

INTERVENTIONS:
Drug: denosumab — subcutaneous injection
  Groups: Men with osteoporosis; Prolia for unapproved indications; Women with post menopausal osteoporosis
Drug: bisphosphonate — The assessment of bisphosphonates includes branded oral bisphosphonates (eg, alendronate [Fosamax®], risedronate [Actonel®], ibandronate [Boniva®/Bonviva®] oral); generic bisphosphonates, including alendronate, neridodronate, and olpadronate; intravenous bisphosphonates including ibandronate IV, and zoledronate [Reclast®/Aclasta®].
  Groups: Women with post menopausal osteoporosis

SUMMARY:
This is a prospective open-cohort study with annual assessment and reporting of descriptive findings from 5 secondary data sources, US Medicare, Optum Research Database (formerly United HealthCare), Scandinavian national health registry databases, including data from Denmark, Sweden, and Norway. The study period will include up to 10 years in each data system depending on data availability. Descriptive statistics will be used to characterize cohorts with respect to patient characteristics and utilization patterns. Person-year adjusted AESI incidence rates will be calculated among postmenopausal women, postmenopausal women with osteoporosis, and exposure cohorts with a final comparative safety analysis. Subsequent sub-studies using US data systems were added to describe men with osteoporosis treated with Prolia and men and women who receive Prolia with glucocorticoid exposure.

DETAILED DESCRIPTION:
This is a prospective open-cohort study with annual assessment and reporting of descriptive findings from 5 secondary data sources, US Medicare,Optum Research Database (formerly United HealthCare), Scandinavian national health registry databases, including data from Denmark, Sweden, and Norway. The study period will include up to 10 years in each data system depending on data availability. Descriptive statistics will be used to characterize exposure cohorts with respect to patient characteristics, clinical features, and AESI risk factors. Person-year adjusted AESI incidence rates will be calculated among postmenopausal women, postmenopausal women with osteoporosis, and exposure cohorts. Exploratory analyses comparing incidence rates of AESI in women with PMO adjusting for potential confounders will also be conducted. Descriptive statistics will be used to characterize denosumab utilisation patterns in patients who receive denosumab for PMO and in subjects who receive Prolia therapy for unapproved indications. Subsequent substudies using US data systems were added to describe men with osteoporosis treated with Prolia and men and women who receive Prolia with glucocorticoid exposure.

ELIGIBILITY:
Criteria: Inclusion Criteria for women with postmenopausal osteoporosis:

* Postmenopausal women: Postmenopausal status will be determined based on age and defined as women ≥ 55 years old. For the Medicare database, only women ≥ 65 years old will be included in the analysis, given that generally all individuals in the US ≥ 65 years old are eligible for Medicare coverage and data on postmenopausal women less than 65 years old will be available for only a small number of women meeting other specialized eligibility criteria.
* Women with Post Menopausal Osteoporosis: The presence of Post Menopausal Osteoporosis will be determined utilizing an algorithm based upon definition of postmenopausal women (≥ 65 years old in Medicare or ≥ 55 years old in other data systems), diagnostic codes indicating osteoporosis, diagnostic codes indicating osteoporotic fracture, and/or relevant postmenopausal osteoporosis treatment codes.
* The inclusion of men and women who have Glucocorticoid Induced Osteoporosis (GIOP) has also been added to the study population. Men and women who receive Prolia with glucocorticoid exposure are included in the ongoing study 20090522 to assess safety in the post-marketing environment

Exclusion Criteria for women with postmenopausal osteoporosis:

• Women with postmenopausal osteoporosis: Women with Paget'sdisease during the 12-month period prior to meeting criteria for inclusion in postmenopausal osteoporosis population will be excluded. Additionally, in US Medicare and United Healthcare, women with a diagnosis of malignancy (excluding non-melanoma skin cancer) or treatment with chemotherapy, hormonal therapy or radiation therapy for cancer up to 12-months before index date will be excluded. In the Scandinavian national registries, women with a diagnosis of cancer according to the patient registry and/or cancer registry up to 12-months prior to meeting criteria for inclusion in postmenopausal osteoporosis population will be excluded.

Inclusion criteria for men with osteoporosis:

• Men ≥ 65 years old in the Medicare database or ≥ 30 years old in andthe Optum Research Database (formerly United HealthCare)United Healthcare who receive at least one denosumab 60 mg injection will be included. All men need to be continuously enrolled for at least 12 months prior to start of follow-up. A diagnosis code of osteoporosis or osteoporotic fracture would not be required because it is known that male osteoporosis is under-diagnosed. The exclusion of patients with cancer or Paget disease (as described in the Exclusion Criteria Section) will ensure that patients treated with Prolia is for osteoporosis but not for other indications. The index date is defined as the date when a patient first satisfies all inclusion criteria.

Exclusion Criteria for men with osteporosis:

* Men with a diagnosis of malignancy (excluding non-melanoma skin cancer) or treatment with chemotherapy, hormonal therapy or radiation therapy for cancer up to 12 months before the index date will be excluded.
* Men with Paget's disease during the 12-month period prior to the index date will also be excluded.

Inclusion criteria for Men and Women Who Receive Prolia With Glucocorticoid Exd Exposure • Men and women identified from Medicare or Optum Research Database who are ≥65 years old (or ≥30 years old in Optum) on or before receiving at least 1 denosumab 60 mg injection or fill after approval date of Prolia for treatment of glucocorticoid-induced osteoporosis (18 May 2018) will be included. This includes both new and prevalent users of denosumab. The index date is defined as the date of the first denosumab administration on or after the approval date fulfilling both the database specific age, 12-month enrollment criteria, and has received a 90-day average daily dose equivalent ≥7.5 mg of prednisone at any time during the previous 12 months.

Exclusion Criteria for Men and Women Who Receive Prolia With Glucocorticoid Exposure

• Men and women with a diagnosis of malignancy (excluding non-melanoma skin cancer) or treatment with chemotherapy, hormonal therapy or radiation therapy for cancer up to 12 months before the index date will be excluded. Men and women with Paget's disease during the 12-month period prior to the index date will also be excluded. The exclusion of subjects with cancer or Paget's disease will ensure that subjects included in the substudy are receiving denosumab for the treatment of osteoporosis, and not for other indications.

Ages: 30 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The main and sub-study populations will be identified based on the following inclusion and exclusion criteria. Patients in Medicare and Optum Research Database (formerly United HealthCare), will need to have appropriate plan coverage to be included in any of the following populations. Appropriate plan coverage for the Optum Research Database (formerly United HealthCare) refers to both pharmacy and medical plan coverage.
  Appropriate plan coverage for the US Medicare database refers to enrollment in traditional fee-for-service Medicare (Medicare Parts A and B coverage and not in a Medicare Advantage plan), plus Part D. The requirement of 12-months of continuous enrollment is not relevant for Scandinavian national registries because all citizens are enrolled in the universal health coverage from birth to death unless they move out of the country.
Sampling Method: Non-Probability Sample
Enrollment: 517991 (Actual)
Dates: Start 2010-05-31 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Incidence rates of Adverse Events of Special Interest (AESI) | Up to 10 years
  Incidence rates of AESI (per 100,000 Person-years) will be assessed in postmenopausal women with osteoporosis (PMO) and by exposure cohort (denosumab or bisphosphonates)
Characteristics and Adverse Events of Special Interest (AESI) risk factors | Up to 10 years
  Describe characteristics, clinical features, and AESI risk factors in women with PMO exposed to denosumab, women with PMO exposed to bisphosphonates, and all women with PMO.
Compare the incidence of the Adverse Events of Special Interests | Up to 10 years
  Compare the incidence of the AESI in women with PMO exposed to denosumab to that in women with PMO exposed to bisphosphonates.
Describe incidence rates of Adverse Events of Special Interest (AESI) | Up to 10 years
  Describe incidence rates of AESI in postmenopausal women.
Describe denosumab utilization patterns | Up to 10 years
  Describe denosumab utilization patterns in patients who receive denosumab therapy for treatment of PMO.
Describe Prolia utilization patterns | Up to 10 years
  Describe Prolia utilization patterns in patients who receive Prolia therapy for unapproved indications (indication, dosage, frequency).

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Xue F, Ma H, Stehman-Breen C, Haller C, Katz L, Wagman RB, Critchlow CW; Denosumab Global Safety Assessment Team. Design and methods of a postmarketing pharmacoepidemiology study assessing long-term safety of Prolia(R) (denosumab) for the treatment of postmenopausal osteoporosis. Pharmacoepidemiol Drug Saf. 2013 Oct;22(10):1107-14. doi: 10.1002/pds.3477. Epub 2013 Jul 15. PMID 23857864
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com